CLINICAL TRIAL: NCT05097131
Title: International Collaboration for Real-World Evidence in Alzheimer's Disease (ICARE AD)- A Prospective Real-World Observational Study of Aducanumab-avwa in Patients With Alzheimer's Disease in the US
Brief Title: An Observational Study of Aducanumab-avwa in Participants With Alzheimer's Disease in the US
Status: Terminated | Type: Observational
Why Stopped: As a result of the national policy for coverage, it is expected there will be limited aducanumab-avwa prescription and usage in routine clinical practice making the study not feasible for enrollment.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-ALZ-11855
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants who have been prescribed with aducanumab-avwa in the post-marketing setting according to standard care of practice will be enrolled.

SUMMARY:
This is a prospective, single-arm, multicenter, non-interventional study of aducanumab-avwa as prescribed in the post-marketing setting in the US. Investigators will be prescribing aducanumab-avwa and participants will be treated according to the standard of care (SoC). Participants will be followed up to 5 years after enrollment and data will be collected at routine visits every 6 to 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a diagnosis of Alzheimer's Disease (AD) and is prescribed aducanumab-avwa by their treating physician.
* Participant's treating physician has made the decision to initiate aducanumab-avwa prior to participant inclusion and independently of the purpose of the study.

Key Exclusion Criteria:

* Participant concurrently participates in any interventional clinical study.
* Participant has ever been treated with aducanumab-avwa at a dose of 3 milligrams per kilogram (mg/kg) or greater prior to signing ICF.
* Participant has ever been treated with aducanumab-avwa and discontinued treatment prior to signing ICF.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been prescribed with aducanumab-avwa in the post-marketing setting according to standard care of practice.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Quick Dementia Rating Scale Informant Version & Patient Version (QDRS-IV/PV) Score | Up to 5 years
  QDRS-IV /PV is rapid dementia staging tool. It is a 10-item questionnaire completed by an informant and a participant. The 10 domains covered are memory and recall, orientation, decision-making and problem-solving abilities, activities outside the home, function at home and hobbies, toileting and personal hygiene, behavior and personality changes, language and communication abilities, mood, and attention and concentration. Each domain is rated on five-point scale with increasing severity of symptoms. Total scores range from 0 to 30 with higher scores representing greater cognitive impairment.
Change from Baseline in Amsterdam Instrumental Activities of Daily Living Questionnaire Short Version (A-IADL-Q-SV) Score | Up to 5 years
  A-IADL-Q-SV is used to measure activities of daily living (ADL) in earliest stages of dementia. It consist of 30 items in 7 categories. All items are rated on a five-point scale, ranging from 'no difficulty' to 'unable to perform'. Scoring is based on item response theory (IRT). A-IADL-Q-SV meet all the basic assumptions of IRT scoring, based on a Graded Response Model: (1) Unidimensionality, which implies that one underlying latent trait determines the items; (2) Local independence, meaning the independence of item responses, conditional on the latent trait; and (3) Monotonicity, meaning the probability of endorsing higher item categories as the trait level increases. The IRT latent trait levels are transformed into a 'T-score' with a range from approximately 20 to 80, a mean of 50 and a standard deviation of 10, with higher 'T-scores' indicating better IADL functioning.
Change from Baseline in Functional Activities Questionnaire (FAQ) Score | Up to 5 years
  FAQ is a 10-item questionnaire designed to assess independence in participants with Alzheimer's Disease by measuring instrumental activities of daily living. Each question is rated on a 4-point Likert scale (0 = normal to 3 = dependent). Total score ranges from 0 to 30 with higher scores indicating more impairment.
Change from Baseline in Montreal Cognitive Assessment Version 8.1 (MoCA v8.1) Score | Up to 5 years
  It is used to detect mild cognitive dysfunction. It assesses 30 items in different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score ranges from 0-30 with lower score indicating poor performance.
Change from Baseline in Neuropsychiatric Inventory Questionnaire (NPI-Q) Score | Baseline up to 5 years
  The NPI-Q assesses twelve behavioral domains common in dementia including; hallucinations, delusions, agitation/aggression, dysphoria/depression, anxiety, irritability, disinhibition, euphoria, apathy, aberrant motor behavior, sleep/night-time behavior change, and appetite/eating change. The questionnaire is given by the clinician to the patient's caregiver who is asked if the behavior described is present in the patient. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale (1 = mild, 2= moderate, and 3= severe) and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale (0 = not distressing at all, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, and 5 = extreme or very severe). The total severity score represents the sum of individual scores and ranges from 0 to 36. The total distress score represents the sum of individual symptom scores and ranges from 0 to 60.
Change from Baseline in Geriatric Depression Scale Short Form (GDS-SF) Score | Up to 5 years
  This is the screening test for depression in elderly people. The questionnaire contains 15 items. Participants indicate the presence or absence of each symptom. The GDS-SF score is the total number of positive depressive items. Score range is from 0-15. Scores of 0-4 are considered normal, 5-8 indicate mild depression, 9-11 indicate moderate depression and 12-15 indicate severe depression.
Change from Baseline in 13-Item Quality of Life in Alzheimer's Disease (QoL-AD) Score | Up to 5 years
  The scale includes 13 items of life domains including the participant's physical health, mood, relationships, activities, and ability to complete tasks. Each item is scored using a scale of 1-4 (poor, fair, good, or excellent). Total score ranges 13-52; higher scores indicate better QOL.
Change from Baseline in Zarit Burden Interview (22-Item) Score | Up to 5 years
  This assesses the level of burden experienced by the principal caregivers of older participants with senile dementia and disabled participants. It consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden.
Change from Baseline in Short Form 12 Version 2 (SF-12v2) Score | Up to 5 years
  It is an alternative to Short Form 36 (SF-36®) for use in large surveys of general and specific populations as well as large longitudinal studies of health outcomes. It consists of eight subscale scores (physical functioning [PF], role-physical [RP], bodily pain [BP], general health [GH], vitality [VT], social functioning [SF], role-emotional [RE], and mental health [MH]). Total score ranges from 0 to 100. Higher scores indicate better health status.
Change from Baseline in Health Care Resource Utilization (HCRU) Using Resource Utilization in Dementia Lite (RUD Lite) | Up to 5 years
  Measures HCRU among older adults with dementia and their caregivers, and time spent on formal and informal care by caregivers. This questionnaire is not scored, it provides information, such as, hospitalizations, time spent assisting with personal ADLs, time spent supervising the participant, social services.
Change form Baseline in Patient Global Impressions Scale of Severity (PGI-S) Score | Up to 5 years
  PGI-S evaluates the severity of participant's condition. PGI -S is a 1-item questionnaire where the response is recorded on a 4-point scale scored as: "normal" (1), "mild" (2), "moderate" (3), or "severe" (4).
Change from Baseline in Patient Global Impression of Change (PGI -C) Score | Up to 5 years
  PGI-C is a 7-point self-administered scale that assesses if there has been a change in the participant's health over time. Participants will rate their change as "1=very much improved," "2=much improved," "3=minimally improved," "4=no change," "5=minimally worse," "6=much worse," or "7=very much worse".

SECONDARY OUTCOMES:
The Number of Participants With Adverse Events (AEs), Including Amyloid-Related Imaging Abnormality (ARIA), andSerious Adverse Events (SAEs) in Aducanumab-avwa-treated Participants in Real-world Per Label Recommendation | Up to 5 years
  An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of amedicinal product, whether or not related to the medicinal product. An SAE is any untoward medical occurrence thatat any dose: results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event) requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent orsignificant disability/incapacity, results in a congenital anomaly/birth defect, is a medically important event.
To Obtain Descriptive Statistics on the Characteristics of the Aducanumab-avwa User Population and on Drug Utilization | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (22):
- United States (22):
  - Research Site, Chula Vista, California
  - Mehdi Meratee MD, Valencia, California
  - Research Site, Boca Raton, Florida
  - Research Site, Bradenton, Florida
  - New Life Medical Research Center, Inc, Hialeah, Florida
  - Miami Jewish Health System, Inc, Miami, Florida
  - Imic, Inc., Palmetto Bay, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Northwest Neurology, Chicago, Illinois
  - Research Site, Ozark, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - South Shore Neurologic Associates, P.A., Patchogue, New York
  - Carolina Clinical Research & Consulting, LLC, Asheboro, North Carolina
  - Research Site, Matthews, North Carolina
  - Research Site, Canton, Ohio
  - Dayton Center for Neurological Associates, Centerville, Ohio
  - Center for Cognitive Health, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Coastal Neurology, PA, Port Royal, South Carolina
  - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - The Memory Clinic, Bennington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/